CLINICAL TRIAL: NCT02125370
Title: Experiences of Pregnant Women Who Use NRT in Pregnancy as Part of a Quit Attempt
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 14024
Record Dates: First submitted 2014-04-23; First posted 2014-04-29 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Qualitative; Nicotine Replacement Therapy; Pregnancy
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nicotine Replacement Therapy
  Interventions: Other: Qualitative and survey

INTERVENTIONS:
Other: Qualitative and survey

SUMMARY:
This study is largely a qualitative study with a small survey component. The aim of the survey would be to gain a quantitative perspective of how women use NRT after this has been prescribed by stop smoking services (SSS). The aim of the qualitative study would be to enhance knowledge of pregnant smoker's views and attitudes about their experiences of using NRT and in particular to understand why pregnant women who start using NRT often discontinue this early or do not use the medication as it is prescribed. This information is important for a number of reasons; firstly it will help health professionals and researchers gain an in depth understanding about how women experience using NRT, which may be used to help devise strategies for encouraging better adherence and which could be used in future clinical trials to gain a clearer understanding as to whether or not NRT is effective in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Quantitative survey;

  * Women who are pregnant
  * Aged 16 or over (no upper age limit)
  * Who have been prescribed NRT (patches/dual therapy) to aid a quit attempt.

Qualitative interview study will include the above plus;

* Women will have used NRT for over 24 hours
* Either not be using NRT as prescribed (as deciphered by the survey questions) or have currently quit NRT (and have either stopped smoking or continue to smoke)

Exclusion Criteria:

* Survey and qualitative interviews

  * Women who cannot understand the study procedure sufficiently in order to provide consent e.g. due to cognitive difficulties
  * Women who are unable to read or understand the consent procedure and study procedures in English.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be identified through two identification sites; New Leaf Stop Smoking Services in Nottinghamshire and Nottingham City. The study will consist of a short survey focussing on how NRT is used during pregnancy. As well as providing information the survey responses will also be able to distinguish who is eligible to participate in qualitative telephone interviews. A subsection of these women will be asked to participate in an interview. The survey and interviews will be conducted as close as possible after participants have had an appointment with a smoking cessation advisor and, have given consent for the researcher to contact them, this is likely to be within a two week period.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
number of women that use NRT after being prescribed | within 4 weeks of taking part in the study
  All women will be asked whether they have used NRT after being given a prescription, this measurement will be obtained within 4 weeks of the participant consenting to take part in the study.

SECONDARY OUTCOMES:
Number of women who adhere to NRT | 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University of Nottingham, Nottingham, Nottinghamshire
  - New Leaf Stop smoking services, Nottingham